CLINICAL TRIAL: NCT03947437
Title: A Phase 1b / 2a, Double-Blind, Randomized, Placebo-Controlled, Antigen Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of LEP-F1 + GLA-SE in Adult Participants in Areas Endemic for Leprosy
Brief Title: Phase 1b/2a Trial to Evaluate LEP-F1 + GLA-SE in Healthy Adults and Leprosy Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Oswaldo Cruz Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASCLIN 002/2020
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Leprosy
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Intervention Model Description: A Phase 1b / 2a, Double-Blind, Randomized, Placebo-Controlled, Antigen Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of LEP-F1 + GLA-SE in Adult Participants in Areas Endemic for Leprosy
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Participants, investigators, study personnel performing any study-related assessments following study injection, and laboratory personnel performing immunology assays will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose (Experimental): 2 μg LEP-F1 + 5 μg GLA-SE will be administered by IM injection on Days 0, 28, and 56 in healthy participants.
  Interventions: Biological: LEP-F1 + GLA-SE
- High dose (Experimental): 10 μg LEP-F1 + 5 μg GLA-SE will be administered by IM injection on Days 0, 28, and 56 in healthy participants.
  Interventions: Biological: LEP-F1 + GLA-SE
- TBD dose in patients (Experimental): TBD μg LEP-F1 + 5 μg GLA-SE will be administered by IM injection on Days 0, 28, and 56 in paucibacillary leprosy patients. Dose will be determined by safety and immunogenicity data from healthy participants.
  Interventions: Biological: LEP-F1 + GLA-SE
- Placebo (Placebo Comparator): Sterile normal saline for injection will be administered by IM injection on Days 0, 28, and 56 in healthy participants and paucibacillary leprosy patients.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LEP-F1 + GLA-SE — Leprosy antigen formulated with an adjuvant.
  Other Names: LepVax
  Arms: High dose; Low dose; TBD dose in patients
Biological: Placebo — Sterile normal saline for injection.
  Arms: Placebo

SUMMARY:
This is a phase 1b/2a, double-blind, randomized, placebo-controlled clinical trial to evaluate the safety, tolerability, and immunogenicity of the LEP-F1 + GLA-SE investigational vaccine compared to placebo.

DETAILED DESCRIPTION:
The proposed clinical trial will establish an initial safety profile for the vaccine in a region endemic for leprosy. The trial will enroll both healthy participants and paucibacillary leprosy patients receiving standard-of-care therapy. Safety at the lower vaccine dose will be demonstrated in healthy participants prior to antigen dose-escalation. Further, safety in all healthy participants will be demonstrated prior to enrolling leprosy patients.

Participants will be randomized within each Group to receive three doses of vaccine or placebo administered IM on Days 0, 28, and 56. Participants will be monitored for one year following the last study injection.

ELIGIBILITY:
Phase 1b

Inclusion Criteria:

1. Men and women between 18 and 55 years old.
2. They should be in good general health, confirmed by a medical history and physical examination, with negative clinical evaluation for leprosy.
3. Female participants of childbearing age should have a negative serum pregnancy test at screening and a negative urine pregnancy test on study vaccination days (D0, D28 and D56). They must not be breast-feeding and are required to use at least one contraceptive method from the time of study inclusion (Day 0) until 30 days after the last injection if they have sex with men.
4. Screening laboratory tests with normal, within laboratory reference limits for:: sodium, potassium, AST, ALT, total bilirubin, alkaline phosphatase, creatinine, glucose, total leukocyte count, hemoglobin and platelet count. Abnormal results may be repeated at the discretion of the Principal Investigator and/or sub-investigators, who may share doubts with the sponsor's Scientific Leader and if necessary with the DSMB.
5. Negative serological tests for: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
6. Normal or not clinically significant urinalysis as determined by the study doctor or designee. Abnormal results may be repeated at the discretion of the Principal Investigator.
7. Must be able to complete the study adverse events diary.
8. Must consent to participate in the study, be able and willing to make all evaluation visits, be accessible by telephone or home visits, and live in the region until study follow-up completion.
9. Having completed the primary vaccination course for Covid 19, at least 14 days before inclusion in the study. If 14 days have not been completed, the participant may be rescheduled for a new eligibility assessment

Exclusion Criteria (Phase 1b)

Individuals who meet ANY of the following criteria will be considered ineligible:

1. History of infection with Mycobacterium leprae.
2. History of exposure to experimental products containing GLA-SE.
3. History of active or documented latent tuberculosis.
4. History of previous infection with other non-tuberculous mycobacteria.
5. Participation in another trial protocol and/or receipt of any trial products in the last 3 months prior to screening.
6. Treatment with immunosuppressive drugs (eg oral or injected steroids, such as prednisone; high doses of inhaled steroids) or cytotoxic therapies (eg chemotherapy or radiation) within 6 months prior to screening.
7. Have received blood transfusion within the last 3 months prior to screening.
8. Donated blood products (platelets, whole blood, plasma, etc.) within the last month prior to screening.
9. Received any vaccine 1 month prior to screening or planned immunizations during the follow-up from D0 to D63 and D154 to D168.
10. History of autoimmune disease or other immunosuppressive causes.
11. History of any other acute or chronic decompensated disease (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, haematological, metabolic or renal disease, uncontrolled hypertension) or use of medication that, in the opinion of the Principal Investigator, may interfere with safety or immunogenicity of the vaccine.
12. Rash, tattoos or any other dermatological condition that may adversely affect the injection site of the vaccine or interfere with its evaluation.
13. Body mass index (BMI) ≥ 32.
14. Systemic arterial hypertension (systolic > 150 or diastolic > 95).
15. History of psychiatric illness with current medication use.
16. Alcohol or drug abuse in the last 6 months prior to screening.
17. Chronic smoker (1 pack or more per day).
18. History of previous anaphylaxis or severe allergic reaction to unknown vaccines or allergens.
19. Individuals who do not wish to cooperate with all procedures recommended in the study protocol.

Inclusion Criteria (Phase 2a)

Participants must meet ALL of the following criteria listed below to be included in the study:

1. Men and women between 18 and 55 years old.
2. Diagnosis of PB leprosy (BI=0) before MDT treatment
3. Female participants of childbearing age should have a negative serum pregnancy test at screening and a negative urine pregnancy test on study vaccination days (D0, D28 and D56). They must not be breast-feeding and are required to use at least one contraceptive method from the time of study inclusion (Day 0) until 30 days after the last injection if they have sex with men.
4. Screening laboratory tests with normal, within laboratory reference limits for: sodium, potassium, AST, ALT, total bilirubin, alkaline phosphatase, creatinine, glucose, total leukocyte count, hemoglobin and platelet count. Abnormal results may be repeated at the discretion of the Principal Investigator and/or sub-investigators, who may share doubts with the sponsor's Scientific Leader and if necessary with the DSMB.
5. Negative serological tests for: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
6. Normal or not clinically significant urinalysis as determined by the study doctor or designee. Abnormal results may be repeated at the discretion of the Principal Investigator.
7. Must be able to complete the study adverse events diary.
8. Must consent to participate in the study, be able and willing to make all evaluation visits, be accessible by telephone or home visits, and live in the region until study follow-up completion.
9. Having completed the primary vaccination course for Covid 19, at least 14 days before inclusion in the study. If 14 days have not been completed, the participant may be rescheduled for a new eligibility assessment

Exclusion Criteria (Phase 2a)

Individuals who meet ANY of the following criteria will be considered ineligible:

1. Previous treatment for leprosy.
2. History of exposure to experimental products containing GLA-SE.
3. History of active or documented latent tuberculosis.
4. History of previous infection with other non-tuberculous mycobacteria.
5. Participation in another trial protocol and/or receipt of any trial products in the last 3 months prior to screening.
6. Treatment with immunosuppressive drugs (eg oral or injected steroids, such as prednisone; high doses of inhaled steroids) or cytotoxic therapies (eg chemotherapy or radiation) within 6 months prior to screening.
7. Have received blood transfusion within the last 3 months prior to screening.
8. Donated blood products (platelets, whole blood, plasma, etc.) within the last month prior to screening.
9. Received any vaccine 1 month prior to screening or planned immunizations during the follow-up from D0 to D63 and D154 to D168.
10. History of autoimmune disease or other immunosuppressive causes.
11. History of any other acute or chronic decompensated disease (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, haematological, metabolic or renal disease, uncontrolled hypertension) or use of medication that, in the opinion of the Principal Investigator, may interfere with safety or immunogenicity of the vaccine.
12. Rash, tattoos or any other dermatological condition that may adversely affect the injection site of the vaccine or interfere with its evaluation.
13. Body mass index (BMI) ≥ 32.
14. Systemic arterial hypertension (systolic > 150 or diastolic > 95).
15. History of psychiatric illness with current medication use.
16. Alcohol or drug abuse in the last 6 months prior to screening.
17. Chronic smoker (1 pack or more per day).
18. History of previous anaphylaxis or severe allergic reaction to unknown vaccines or allergens.
19. Individuals who do not wish to cooperate with all procedures recommended in the study protocol.

Vital signs are performed after participants have sat for five minutes without hot or cold drinks or smoking for the past five minutes. Vital signs can be performed up to three times to allow resolution of transient conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1b_The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection. | 7 days following each injection
  The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection.
Phase 1b_Number of participants experiencing unsolicited AEs | Days 0 to 84
  The number of participants spontaneously reporting adverse events from Day 0 to Day 84.
Phase 1b_The number of adverse events attended by physicians considered related to any of the study injections reported at any time during the study period. | Days 0 to 421
  The number of adverse events attended by physicians considered related to any of the study injections reported at any time during the study period.
Phase 1b_The LEP-F1 specific T cell IFN--γ production responses in assay with PBMCs evaluated by ELISA on Days 0, 35 and 63. | Days 0, 35 and 63.
  The LEP-F1 specific T cell IFN-γ production responses in assay with PBMCs evaluated by ELISA on Days 0, 35 and 63.
Phase 2a_The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection. | 7 days following each injection
  The number of participants who receive the injection and experience local and systemic reactions within 7 days of each study injection.
Phase 2a_The number of participants spontaneously reporting adverse events from Day 0 to Day 84. | Day 0 to Day 84.
  The number of participants spontaneously reporting adverse events from Day 0 to Day 84.
Phase 2a_The number of physician-assisted adverse events considered related to any of the study injections reported at any time during the study period | Day 0 to Day 421
  The number of physician-assisted adverse events considered related to any of the study injections reported at any time during the study period
Phase 2a_The frequency and intensity of solicited adverse events within 7 days of each study injection. | 7 days following each injection
  The frequency and intensity of solicited adverse events within 7 days of each study injection.
Phase 2a_The frequency and intensity of unsolicited adverse events during study participation (D0 to D421). | Day 0 to Day 421
  The frequency and intensity of unsolicited adverse events during study participation (D0 to D421).
Phase 2a_The frequency and causality of serious adverse events occurring during study participation (D0 to D421). | Day 0 to Day 421
  The frequency and causality of serious adverse events occurring during study participation (D0 to D421).

SECONDARY OUTCOMES:
Phase 1b_IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63, and 168. | Days 0, 35, and 63
  IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63, and 168
Phase 1b_ The T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0, 35, 63, and 168.whole blood assay | Days 0, 35, 63 and 168
  The T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0, 35, 63, and 168.
Phase 2a_IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63, and 168. | Days 0, 35, 63, and 168.
  IgG antibody responses to LEP-F1 by ELISA on Days 0, 35, 63, and 168.
Phase 2a_T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0, 35, 63, and 168. | on Days 0, 35, 63, and 168.
  T cell responses measured by LEP-F1-specific cytokine production in PBMC assay by ELISA or multiplex assay on Days 0, 35, 63, and 168.
Phase 2a_The neurological nerve function as measured by clinical and neurophysiological tests | Day 0 to Day 421
  The neurological nerve function as measured by clinical and neurophysiological tests
Phase 2a_The number of participants who received LepVax and had episodes of RR after the start of the study. | Day 0 to Day 421
  The number of participants who received LepVax and had episodes of RR after the start of the study.
Phase 2a_The number of M. leprae genome copies (bacillus quantification). | Day 0 to Day 421
  The number of M. leprae genome copies (bacillus quantification).

OTHER OUTCOMES:
Phase 1b_The T cell responses measured by intracellular cytokine (ICS) staining in PBMCs on Days 0, 35, 63, and 168. | Days 0, 35, 63, and 168.
  The T cell responses measured by intracellular cytokine (ICS) staining in PBMCs on Days 0, 35, 63, and 168.
Phase 1b_The assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay. | Day 0 and 163
  The assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay.
Phase 2a_The T cell responses measured by intracellular cytokine staining of PBMCs on Days 0, 35, 63 and 168 | Days 0, 35, 63 and 168
  The T cell responses measured by intracellular cytokine staining of PBMCs on Days 0, 35, 63 and 168
Phase 2a_The Assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay | Day 0 and 63
  The Assays of candidate biomarkers measured on Day 0 and 63 including gene expression signatures and serum protein multiplex assay

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Schmitz Pereira, PHD, Principal Investigator — Instituto Oswaldo Cruz
Locations (1):
- Veronica Schmitz Pereira, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No